CLINICAL TRIAL: NCT05991557
Title: Peroneus Longus Autograft Use in Knee, Shoulder, Elbow Ligaments Reconstruction Surgery : Effect On Ankle And Foot Function
Brief Title: Peroneus Longus Graft :Effect in Foot and Ankle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Sabra Ahmed, resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: peroneus longus graft
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Ligament Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): peroneus longus autograft
  Interventions: Procedure: peroneus longus autograft

INTERVENTIONS:
Procedure: peroneus longus autograft — Peroneus longus tendon graft will be harvested with a longitudinal skin incision at 2 to 3 cm (2 finger-breadths) above and 1 cm (1 finger-breadth) behind the lateral malleolus, followed by superficial fascia incision in line with skin incision followed by incision of the tendon sheath proximal to the retinaculum. The peroneus longus and peroneus brevis tendons will be then identified. The tendon division location marked at 2 to 3 cm above the level of the lateral malleolus.The peroneus longus tendon will be exposed on its posterolateral surface through the incision after carefully incising the fascia

SUMMARY:
The purpose of this study is to report the ankle and foot functions via American orthopedic foot and ankle society score (AOFAS), peronei muscle testing ,handheld dynamometer and radiological outcomes after harvesting autogenous peroneus longus tendons for ligaments reconstruction.

DETAILED DESCRIPTION:
Using a Peroneus longus tendon (PLT) as an autograft is a common procedure and has been used previously for deltoid ligament reconstruction in flatfoot deformity correction . Recently, (PLT) is gaining popularity as a graft option in primary anterior cruciate ligament (ACL) reconstruction surgeries with biomechanical studies showing tensile strength and clinical outcomes comparable to quadrupled hamstring grafts.

In addition to using PLT for isolated (ACL), it is also used in posterior cruciate ligament (PCL) reconstruction, medial collateral ligament reconstruction, posterolateral corner reconstruction of the knee, or knee multiple ligament injuries . The partial-thickness of the tendon has been used variably in knee ligament surgery..

Being a powerful muscle in plantar flexion and eversion of the foot, there might be associated ankle functional impairment. To the authors knowledge, there is a gap in science evaluating donor site morbidity. The aim of this study is to report the clinical and functional outcome of the donor site for better explanation of the cons and pros of using PLT as a graft in joint ligamentous injury .

ELIGIBILITY:
Inclusion Criteria:

1. clinical and radiological diaginsis of joint ligament injury and needs to ligament reconstruction .
2. people with asymptomatic ankle and foot pre and post injury

Exclusion Criteria:

1. Associated ankle and/or foot fractures.
2. Associated hip or pelvic fractures
3. Abnormal ankle function pre-injury.
4. Contralateral limb fractures
5. Traumatic brain injury (TBI) that limits their ability to participate in their post-operative care;
6. Presence of neurological condition that result in spasticity or any abnormal lower limb muscles tone.
7. Any condition that would preclude the ability to comply with post-operative guidelines.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
peronei muscle strength testing using handheld dynamometer | preoperative, three months postoperative and six months postoperative
  power of plantar flexion and eversion of foot and ankle

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 2- Rudy ME, Phatama KY (2017) Tensile strength comparison between peroneus longus and hamstring tendons: a biomechanical study. Int J Surg Open 9:41-44 — http://doi.org/10.1016/j.ijso.2017.10.002
- See also: Shi F-D, Hess DE, Zuo J-Z et al (2019) Peroneus longus tendon autograft is a safe and effective alternative for anterior cruciate ligament reconstruction. J Knee Surg 32:804-811 — http://doi.org/10.1055/s-0038-1669951
- See also: -Setyawan R, Soekarno NR, Asikin AIZ, Rhatomy S (2019) Posterior cruciate ligament reconstruction with peroneus longus tendon graft: 2-years follow-up. Ann Med Surg 43:38-43 — http://doi.org/10.1016/j.amsu.2019.05.009